CLINICAL TRIAL: NCT00152984
Title: A 12-week Randomised, Double Blind, Placebo Controlled, Parallel Group Trial Evaluating the Efficacy and Safety of Inhaled Tiotropium 18μg q.d. in Patients With COPD and a Concomitant Diagnosis of Asthma
Brief Title: Efficacy and Safety of Tiotropium in Patients With COPD and Concomitant Diagnosis of Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.301
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

INTERVENTIONS:
Drug: Tiotropium inhalation capsules
Drug: Placebo inhalation capsules

SUMMARY:
The primary objective of this study is to demonstrate the superiority of tiotropium compared to placebo in the treatment of patients with COPD and a concomitant diagnosis of asthma

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD and diagnosis of asthma before the age of 30
* Current or ex-smokers with a cigarette smoking history of at least 10 pack-years
* Treatment with inhaled steroids at least 1 year before study entry
* FEV1 increase of more than 12% 30 min. after 400 mcg salbutamol or documented reversibility of 12% documented during the past 5 years
* FEV1 increase of more than 200 mL 30 min. after 400 mcg salbutamol or documented increase of 200 mL after reversibility test within the last 5 years
* Post bronchodilator FEV1 less than 80% predicted normal (ECCS) at visit 1
* Post bronchodilator FEV1 less than 70% of FVC at visit 1

Exclusion criteria:

* Respiratory infection or exacerbation 6 weeks prior to Visit 1 or during run-in period.
* Significant diseases other than COPD or asthma
* Myocardial infarction within the last 6 months
* Unstable or life-threatening cardiac arrhythmia requiring intervention or change in therapy in the last year
* Hospitalisation for heart failure (NYHA Class III or IV) within the last year
* History of life-threatening pulmonary obstruction, cystic fibrosis or clinically evident bronchiectasis
* Known active tuberculosis
* History of thoracotomy with pulmonary resection
* History of cancer within the last 5 years (excluding treated basal cell carcinoma)
* Patients requiring oxygen therapy for more than 1 hour per day
* Patients currently in a pulmonary rehabilitation programme or who have completed such a programme within 4 weeks before Visit 1
* Known hypersensitivity to anticholinergic drugs or lactose

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472
Dates: Start 2004-12; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
AUC(0-6) FEV1 (Area under the curve of change in FEV1 from baseline to 6 hours post dose) | after 12 weeks of treatment

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 12 weeks
Peak expiratory flow rate (PEFR) | 12 weeks
Use of rescue medication | 12 weeks
AUC0-6hFEV1 | after first dose on Day 1 and after 4 weeks of treatment
Change in trough FEV1 (i.e. trough response) from baseline. | after 4 and 12 weeks of treatment
Change in peak FEV1 from baseline (=peak response) after first dose | after 4 and 12 weeks of treatment
AUC0-6hFVC defined in the same way as for FEV1. | Day 1, week 4
Trough FVC defined in the same way as for FEV1. | Day 1, week 4
Peak FVC defined in the same way as for FEV1 | Day 1, week 4
Weekly average PEFR in the morning (a.m. pre-dose measurement) and in the evening (p.m. measurement). | 12 weeks
Weekly average number of puffs of rescue medication used | 12 weeks
Occurrence of adverse events | 12 weeks
Change from baseline in pulse rate and systolic and diastolic blood pressure (seated) measured just before spirometry | 12 weeks
Change from baseline in Physical examination | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (65):
- Belgium (7):
  - CHU Sart Tilman, Angleur
  - A.Z. VUB, Brussels
  - Boehringer Ingelheim Investigational Site, Genk
  - Boehringer Ingelheim Investigational Site, Hasselt
  - St. Elisabethziekenhuis, Herentals
  - Clinique Reine Astrid, Malmedy
  - Sint-Elisabethziekenhuis, Turnhout
- Canada (9):
  - VGH Research Pavillion, Vancouver, British Columbia
  - BG 034, Room C2027, Winnipeg, Manitoba
  - Department of Medicine, Health Sciences Centre, Hamilton, Ontario
  - Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Respiratory Research Lab, Toronto, Ontario
  - Department of Respiratory Medicine, Toronto, Ontario
  - Centre de Recherche Clinique -CUSE, Sherbrooke, Quebec
  - Hopital Laval, Ste-Foy, Quebec
- Denmark (6):
  - Lungemedicinsk Forskning 2B, Aarhus
  - Lungemedicinsk afdeling Y, Hellerup
  - Medicinsk afdeling B0642, Hiller?d
  - Lungemedicinsk Klinik, Hvidovre
  - H:S Bispebjerg Hospital, K?benhavn NV
  - Lungemedicinsk Forskning, Odense C
- France (12):
  - Hopital d'Annecy, Annecy
  - Hopital Prive Antony, Antony
  - Boehringer Ingelheim Investigational Site, Chamalières
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital Ambroise Pare, Marseille
  - Hopital Notre Dame de Bon Secours, Metz
  - Boehringer Ingelheim Investigational Site, Montpellier
  - Hopital Arnaud de Villeneuve, Montpellier
  - Boehringer Ingelheim Investigational Site, Nantes
  - Centre Medical Erdre St Augustin, Nantes
  - Boehringer Ingelheim Investigational Site, Nice
  - Hopital Maison blanche, Reims
- Germany (13):
  - Boehringer Ingelheim Investigational Site, Berlin
  - MEDARS GmbH, Berlin
  - Boehringer Ingelheim Investigational Site, Bonn
  - Med. Einrichtung der Universitat zu Koln, Cologne
  - Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Fürth
  - Inamed Research GmbH & Co. KG, Gauting
  - Boehringer Ingelheim Investigational Site, Gelnhausen
  - ClinPharm Internat. GmbH & Co. KG, Görlitz
  - Pneumologisches Forschungsinstitut GmbH am Krankenhaus, Hamburg
  - Boehringer Ingelheim Investigational Site, Minden
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Rüdersdorf
- Italy (4):
  - A. O. Universitaria di Ferrara - Arcispedale S. Anna, Ferrara
  - A.O. S. Martino e Cliniche Universitarie di Genova, Genova
  - Universita di Genova, Genova
  - A.O. Pisana, Pisa
- Netherlands (7):
  - Ziekenhuisgroep Twent, Almelo
  - Amphia ziekenhuis, Breda
  - Atrium medisch centrum, Heerlen
  - Ziekenhuigroep Twente, Hengelo
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Antonius Ziekenhuis, Sneek
  - Maxima Medisch Centrum, Velthoven
- South Africa (7):
  - Boehringer Ingelheim Investigational Site, Bellville
  - Boehringer Ingelheim Investigational Site, Cape Town
  - Boehringer Ingelheim Investigational Site, Durban
  - Boehringer Ingelheim Investigational Site, George
  - Boehringer Ingelheim Investigational Site, Paarl
  - Boehringer Ingelheim Investigational Site, Pretoria
  - Boehringer Ingelheim Investigational Site, Somerset West

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/17920256